CLINICAL TRIAL: NCT04192877
Title: Validation and Inter-rater Reliability of the Vagus Nerve Neurodynamic Test Among Healthy Subjects.
Brief Title: Validity and Inter-rater Reliability fo the Vagus Nerve Neurodynamic Test Among Healthy Subjects
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Giacomo Carta, Principal Investigator, Clinical Professor, University of Turin, Italy
Other Study IDs: 139870-14/03/2019
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Vagus Nerve Diseases; Diagnoses Disease
Keywords: Validation Studies; Vagus Nerve Diseases; Diagnostic imaging; Motion analysis; Healthy Volunteers
MeSH Terms: conditions — Vagus Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: 30 healthy subjects from both genders, aged between 18 and 60 years will be screened for neurological deficits. If neurological examination will be negative markers for motion capture, analysis will be placed on the chest and shoulders and a rubber band, with 3 markers, will be placed on the forehead. The subjects will be invited to lay on a medical table and heart rate (HR) will be assessed at rest. The vagus nerve neurodynamic test (VN-NDT) will be performed by an expert and a novice, in a random order, and under ultrasound imaging (USI). Assessors will be blinded to their results. Heart rate (HR) of the subjects will be monitored and a pain drawaing tools will be used to describe and locate the symptoms induced during the test administration.
  Interventions: Diagnostic Test: Vagus Nerve Neurodynamic test

INTERVENTIONS:
Diagnostic Test: Vagus Nerve Neurodynamic test — The VN-NDT has been developed starting from the VN morphology selecting the physiological movements that induce the greater mechanical tension on the nerve. The subjects will be assessed supine on an examination table with assessors standing at the cranial short side of the table. Upper cervical flexion and contralateral lateral flexion had been selected for loading the intracranial portion. The ipsilateral neck rotation had been selected for loading the cervical tract. Keeping the subject's head in the final movements combination gentle movements of the upper abdomen caudally and cranially had been selected for loading the thoracic tract and used as discrimination maneuver. The test will be declared positive (indicating abnormal responses) if symptoms will be felt in anatomical regions other than the neck on the same side of the test and discrimination maneuvers changed the subject's symptoms indicating a neurogenic source, otherwise it will be declared negative.
  Other Names: Heart rate monitoring using a digital pulsossimeter

SUMMARY:
Vagus nerve neurodynamic test (VN-NDT) will be validated detecting the changes in vagus nerve anatomical position due to the combination of movements of the test. Healthy subjects will be enrolled and screened for neurological problems. A checklist for autonomic dysfuntion symptoms will be administered and heart rate at rest will be measured. Inter-rater reliability will be assessed comparing positive and negative cases identified by two blinded assessors, one expert and one novice. It will also be monitored and compared the amount of motion induced by the expert and the novice assessors during the VN-NDT admimistration. If symptoms will be produced by the VN-NDT using a pain drawing tool it will be defined the qualitiy and the location of them. Accuracy of the VN-NDT will be tested in the autonomic dysfunction symptom detection.

DETAILED DESCRIPTION:
_A growing body of evidence has shown that the Vagus Nerve (VN) is not only the main anatomical structure responsible for the brain and guts communication but is also a target for many interventions in which drugs or classic treatments have failed. The VN cervical tract stimulation has reported positive results for high social burden problems like acute and chronic pain, psychiatric diseases, disturbs of consciousness and epilepsy. Also, it is well known that the selective tension of the Peripheral Nervous System, or neurodynamic test (NDT), is useful for diagnosis and treatment of neuropathic diseases and pain. Over the last 30 years NDTs were validated for upper and lower limb nerves but nowadays a VN-NDT is lacking and could be a potential alternative in diagnosis and treatment for critical or neglected conditions. Methods_ An estimated sample of 30 healthy participants will complete a questionnaire on vagal symptoms and perceived health status. A neurological assessment of the cervical tract will be performed before the test. The VN-NDT will be administered through a standardized sequence of physiological neck movements. Symptoms and heart rate (HR) will be monitored. Validity of NDT will be tested with ultrasonography assessment (C6-VN distance) during the tests administered by an expert and a novice. Motion of both assessors and subjects will be tracked through an infra-red optoelectronic system. Inter-examiner accordance will be obtained and comparisons between assessors' positive and negative tests due to symptoms provocation and reduction (Cohen's Kappa) will be performed. A two-way analysis of variance (ANOVA) will be performed with factors experience and side tested (2 × 2). Receiver operating characteristic (ROC) curves will be adopted to define the accuracy, sensitivity, specificity, positive and negative likelihood ratios of the VN-NDT in autonomic dysfunction symptoms detection and on perceived health status.Results_ It is expected to determine the inter-examiner accordance and to not detect significant assessors effects on test results. It is also expected to detect a change of the C6-VN distance and HR during the test and to estimate the accuracy of the test for autonomic dysfunctions detection.Conclusions_ Normative physiological values parameter variations at the administration of the VN-NDT are fundamental to determine the hallmarks needed to screen clinical and preclinical conditions involving autonomic dysfunctions_

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 70 years old
* Subjects that have signed the written informed consent

Exclusion Criteria:

* Subjects with significant neck pain or headache (with NRS greater than 3/10)
* Pregnancy
* Recent neck surgery or significant trauma in the preceding 3 months
* Cancer or inflammatory disorders spinal cord or cauda equina signs
* Widespread neurological disorders affecting the tone of upper limb and neck muscles
* Underlying diseases, such as diabetes mellitus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects that want to participate in the study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Vagus nerve neurodynamic test (VN-NDT) | The test will be administered twice for each side, once by an expert and once by a novice.
  combination of physiological movements of the neck (upper cervical flexion, contralateral lateral flexion, ipsilteral rotation and gentle movements of the upper abdomen caudally and cranially to increase tension on the thoracic tract of the VN)
Ultrasound imaging (USI) | USI will be administered twice for each side, once by an expert and once by a novice.
  Axial scans will be obtained using the inferior margin of the thyroid as initial reference from which the probe will be moved laterally to the region of the transverse processes. The probe will also be moved cranially till anterior tubercle of C6 detection. Distance between VN and C6 anterior tubercle will be measured at rest and at the final position of the VN-NDT to quantify the lateralization or proximalization of the VN induced by the test.
Motion capture analysis (MCA) | MCA will be used for the duration the VN-NDT administered twice for each side, once by an expert and once by a novice.
  Throughout the whole duration of VN-NDT with real-time USI assessment, the three-dimensional head orientation of the subjects will be recorded at 100 Hz by means of an optoelectronic motion capture system (Smart-DX, BTS S.p.A., Milano, Italy). A cluster with three retroreflective markers (diameter: 15 mm) will be secured on the subject's head using an elastic band; three additional markers will be fixed on the acromia and on the sternum. The time event corresponding to the obtainment of a proper USI in the rest and final head positions will be manually annotated upon explicit communication by the USI operator.System calibration will be conducted according to the manufacturers' guidelines and returned an average error in marker position of 0.35 mm, on a working volume of 2.6 x 1.8 x 2.5 m3
Short-term autonomic response (STAR) | HR will be measured at rest and end of the VN-NDT for each sides (4 times by an expert and 4 times by a novice).
  The heart rate will be taken (HR) as reference comparing the HR from rest to the HR keeping the head and neck of the subjects in the end position of the VN-NDT for 5 seconds

SECONDARY OUTCOMES:
Checklist for symptoms related to autonomic peripheral neuropathy (APN) and VN dysfunction | The checklist will be administred once. Before the neurological examination
  A checklist for the presence of any symptoms and signs reported in literature to be linked with APN and VN diseases was fulfilled by every participant (Orthostatic Hypotension; Nausea; Digestion Alterations; Breathing Alterations (shortness of breath); Voice Changes; Altered deglutition; Perceived augmented HR;Perceived reduced HR; Burning sensation in the stomach; Constipation; Diarrheal; Vomit; Augmented lacrimation; Reduced lacrimation; Augmented salivation; Reduced salivation; Head and neck sweating attacks; Head and neck skin dryness; Sleep alteration)
Perceived health status (PHS) | The PHS will be administred once. Before the neurological examination
  A 11 point Likert scale was administered to assess the Perceived health status (100 the best 0 the worst health status ever)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, Msc, Principal Investigator — University of Turin, Italy
Locations (1):
- Movement and Posture Analysis Lab, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All of the individual particiapnt data collected during the trial will be shared after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following the publication. No end date.
Access Criteria: Anyone who wishes to access the data.
URL: http://www.mendeley.com/profiles/giacomo-carta/

REFERENCES:
- [Derived] Carta G, Seregni A, Casamassima A, Galli M, Geuna S, Pagliaro P, Zago M. Validation and Reliability of a Novel Vagus Nerve Neurodynamic Test and Its Effects on Heart Rate in Healthy Subjects: Little Differences Between Sexes. Front Neurosci. 2021 Sep 6;15:698470. doi: 10.3389/fnins.2021.698470. eCollection 2021. PMID 34552462